CLINICAL TRIAL: NCT00914927
Title: A Phase 2, Randomized, Multicenter, Placebo-Controlled, Double-Blind, Parallel-Group Study to Evaluate the Efficacy, Safety, and Population Pharmacokinetics of Once-Daily Oral E5501 Tablets Used Up to 7 Days in Subjects With Chronic Liver Diseases and Thrombocytopenia Prior to Elective Surgical or Diagnostic Procedures
Brief Title: Once-Daily Oral Avatrombopag Tablets Used in Subjects With Chronic Liver Diseases and Thrombocytopenia Prior to Elective Surgical or Diagnostic Procedures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E5501-G000-202
Record Dates: First submitted 2009-06-04; First posted 2009-06-05 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Thrombocytopenia Related to Chronic Liver Disease
Keywords: Thrombocytopenia; chronic liver disease
MeSH Terms: conditions — Thrombocytopenia | interventions — avatrombopag

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Avatrombopag
- 2 (Experimental)
  Interventions: Drug: Avatrombopag; Drug: Placebo
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Avatrombopag — Avatrombopag first Dose 80 mg followed by 10 mg a day for up to 6 additional days
  Arms: 1
Drug: Avatrombopag — Avatrombopag first Dose 80 mg followed by 20 mg a day for 3 days and then Placebo for 3 additional days
  Arms: 2
Drug: Placebo — Placebo or inactive substance once a day for up to 7 days
  Arms: 2; 3

SUMMARY:
The purpose of this study is to evaluate the efficacy of once-daily Oral avatrombopagin subjects with chronic liver diseases and thrombocytopenia prior to elective surgical or diagnostic procedures, to evaluate the safety of short-term administration of avatrombopag and to evaluate the pharmacokinetics (PK) of E5501.

ELIGIBILITY:
Key Inclusion Criteria:

1. Males or females ≥ 18 years of age
2. Thrombocytopenia (defined as a platelet count ≥ 10,000 - ≤ 50,000 (+15%)/mm^3 )
3. Model for End-Stage Liver Disease (MELD) scores ≤ 24
4. Chronic liver diseases due to one of the following three etiologies:

   Chronic Viral Hepatitis from one of the following categories
   * Chronic Hepatitis C (defined as the presence of anti-hepatitis C virus [HCV] antibodies and/or detectable serum HCV ribonucleic acid [RNA] levels)
   * OR chronic Hepatitis B (defined as the presence of hepatitis B surface antigen [HBsAg] and/or detectable serum hepatitis B virus [HBV] deoxyribonucleic acid [DNA])
   * OR chronic Hepatitis B and C co-infection (as defined by the above bullet points)
   * OR chronic Hepatitis C and history of alcohol abuse
   * OR chronic Hepatitis B and history of alcohol abuse

   NASH diagnosed as:
   * absence of serologic evidence of viral hepatitis and
   * convincing evidence of a history of minimal or no alcohol consumption, and
   * histologic picture of steatohepatitis OR
   * when histology is unavailable, then clinical, radiographic and laboratory evidence of NASH

   Alcoholic liver disease diagnosed as:
   * absence of serologic evidence of viral hepatitis and
   * history of heavy alcohol consumption and
   * histologic picture of alcoholic liver disease OR
   * when histology is unavailable, then clinical, radiographic and laboratory evidence of hepatitis combined with years of excessive alcohol intake
5. Subjects who are scheduled to undergo an elective invasive procedure between 1 to 4 days post last dose of study drug.
6. Adequate renal function as evidenced by a calculated creatinine clearance ≥50 mL/minute per the Cockcroft and Gault formula
7. Life expectancy ≥3 months

Key Exclusion Criteria:

1. Hepatic encephalopathy that cannot be effectively treated.
2. Platelet transfusion within 7 days prior to the first dose of study drug
3. Received blood products, eg, FFP and cryoprecipitate 7 days prior to the first dose of study drug
4. Have surgical or diagnostic procedure scheduled during the Randomization Phase (Day 1 to Day 8) of this study
5. Interferon use within 2 weeks of Day 1
6. Hormonal contraceptive use within 60 days of study entry
7. History of human immunodeficiency virus (HIV) infection
8. Any prohibited concomitant medications or therapy that cannot be discontinued by Visit 1
9. Active alcohol abuse, active alcohol dependence syndrome, drug abuse, or drug dependence within 6 months of the study start (unless participating in a controlled rehabilitation program)
10. Acute alcoholic hepatitis (chronic alcoholic hepatitis is allowed) within 6 months of the study start
11. History of any primary hematologic disorder
12. History of arterial or venous thrombosis, including thrombosis of any part of the splenic-mesenteric system
13. Any evidence of current portal vein thrombosis (PVT) as detected by Doppler sonography or appropriate MRI/CT imaging at Screening and/or within approximately 30 days prior to Screening
14. Any acute/active bleeding (gastrointestinal [GI], central nervous system [CNS], etc)
15. Uncompensated congestive heart failure (New York Heart Association [NYHA] Class III or IV)
16. Pre-diagnosed Immune Thrombocytopenic Purpura (ITP)
17. History of Myelodysplastic Syndrome (MDS)
18. Females who are pregnant (positive β-hCG test ) or breastfeeding
19. Current use of recreational drugs
20. Post-transplant patients
21. Subjects who have participated in another investigational trial within 30 days prior to Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2009-05; Primary Completion 2011-11-11 (Actual); Study Completion 2011-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Jenkins, Study Director — Eisai Inc.
Locations (1):
- Ochsner Clinic Foundation, New Orleans, Louisiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: 20 mg Avatrombopag, 1G Formulation: Participants received a 100 mg loading dose of the first generation (1G) formulation avatrombopag on Day 1, followed by 20 mg of the 1G formulation avatrombopag once daily on Days 2 to 7.
- Cohort A: 40 mg Avatrombopag, 1G Formulation: Participants received a 100 mg loading dose of the 1G formulation avatrombopag on Day 1, followed by 40 mg of the 1G formulation avatrombopag once daily on Days 2 to 7.
- Cohort A: 80 mg Avatrombopag, 1G Formulation: Participants received a 100 mg loading dose of the 1G formulation avatrombopag on Day 1, followed by 80 mg of the 1G formulation avatrombopag once daily on Days 2 to 7.
- Cohort A: Placebo, 1G Formulation: Participants received the 1G formulation avatrombopag-matched placebo loading dose on Day 1, then once daily on Days 2 to 7.
- Cohort B: 0 mg Avatrombopag, 2G Formulation: Participants received an 80 mg loading dose of the second generation (2G) formulation avatrombopag on Day 1, followed by 10 mg 2G formulation avatrombopag once daily on Days 2 to 7.
- Cohort B: 20 mg Avatrombopag, 2G Formulation: Participants received an 80 mg loading dose of the 2G formulation avatrombopag on Day 1, followed by 20 mg 2G formulation avatrombopag once daily on Days 2 to 4 followed by 2G avatrombopag-matched placebo once daily on Days 5 to 7.
- Cohort B: Placebo, 2G Formulation: Participants received the 2G formulation avatrombopag-matched placebo loading dose on Day 1, then once daily on Days 2 to 7.
Period: Overall Study
Arm/Group | Cohort A: 20 mg Avatrombopag, 1G Formulation | Cohort A: 40 mg Avatrombopag, 1G Formulation | Cohort A: 80 mg Avatrombopag, 1G Formulation | Cohort A: Placebo, 1G Formulation | Cohort B: 0 mg Avatrombopag, 2G Formulation | Cohort B: 20 mg Avatrombopag, 2G Formulation | Cohort B: Placebo, 2G Formulation
Started | 18 | 16 | 17 | 16 | 21 | 21 | 21
Completed | 16 | 14 | 17 | 14 | 19 | 21 | 21
Not Completed | 2 | 2 | 0 | 2 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Administrative/Other | 2 | 1 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) population included all participants who were randomized into the study, received study medication, and had a post-treatment assessment.
Groups:
- Cohort B: 10 mg Avatrombopag, 2G Formulation: Participants received an 80 mg loading dose of the second generation (2G) formulation avatrombopag on Day 1, followed by 10 mg 2G formulation avatrombopag once daily on Days 2 to 7.
- Total: Total of all reporting groups
Arm/Group | Cohort A: 20 mg Avatrombopag, 1G Formulation | Cohort A: 40 mg Avatrombopag, 1G Formulation | Cohort A: 80 mg Avatrombopag, 1G Formulation | Cohort A: Placebo, 1G Formulation | Cohort B: 10 mg Avatrombopag, 2G Formulation | Cohort B: 20 mg Avatrombopag, 2G Formulation | Cohort B: Placebo, 2G Formulation | Total
Number analyzed (Participants) | 18 | 16 | 17 | 16 | 21 | 21 | 21 | 130
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.3 (7.16) | 52.8 (7.78) | 55.2 (5.96) | 54.2 (6.87) | 53.9 (5.48) | 56.8 (6.46) | 55.6 (6.52) | 54.8 (6.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 6 | 5 | 10 | 7 | 7 | 42
  Male | 14 | 13 | 11 | 11 | 11 | 14 | 14 | 88

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Response
Description: Platelet counts (PC) were determined from blood draws. A responder is defined as a participant having an increase of at least 20,000/mm^3 PC from Baseline and a PC greater than 50,000/mm^3 at least once during Day 4 through Day 8. Missing PC assessments at any given time point was considered to be a non-response at that point and were not estimated. For PC measurements taken after the last dose day (end of treatment (EOT)), the postdose windows applied. If there was more than one PC within the same analysis visit window, the following selection rules were applied sequentially to determine which PC was used for that time point: 1) the PC that was closer to the target date was used, 2) if PC were equal-distance in days from the target day, the later one based on measurement date and time was used, and 3) if there was more than one PC on the same day, if it was a baseline record, the largest one was used; if it was a postbaseline record, the smallest one was used.
Time Frame: Day 8 (Visit 5, EOT)
Population: Intent-to-treat (ITT) population included all participants who were randomized into the study, received study medication, and had a posttreatment assessment. The ITT population was analyzed as randomized.
Measure: Number; unit: Percentage of participants
Groups:
- Cohort A: 40 mg Avatrombopag , 1G Formulation: Participants received a 100 mg loading dose of the 1G formulation avatrombopag on Day 1, followed by 40 mg of the 1G formulation avatrombopag once daily on Days 2 to 7.
- Cohort B:10 mg Avatrombopag, 2G Formulation: Participants received the 1G formulation avatrombopag-matched placebo loading dose on Day 1, then once daily on Days 2 to 7.
Arm/Group | Cohort A: 20 mg Avatrombopag, 1G Formulation | Cohort A: 40 mg Avatrombopag , 1G Formulation | Cohort A: 80 mg Avatrombopag, 1G Formulation | Cohort A: Placebo, 1G Formulation | Cohort B:10 mg Avatrombopag, 2G Formulation | Cohort B: 20 mg Avatrombopag, 2G Formulation | Cohort B: Placebo, 2G Formulation
Number analyzed (Participants) | 18 | 16 | 17 | 16 | 21 | 21 | 21
Percentage of participants
  Yes response | 38.9 | 31.3 | 76.5 | 6.3 | 42.9 | 52.4 | 9.5
  No response | 61.1 | 68.8 | 23.5 | 93.8 | 57.1 | 47.6 | 90.5

2. Secondary Outcome: Change in Platelet Count on Day 8 (Visit 5 and/or End of Treatment) From Baseline
Description: Platelet counts were determined from blood draws. Missing PC assessments at any given time point was considered to be a non-response at that point and were not estimated. For PC measurements taken after the last dose day (EOT), the postdose windows applied. If there was more than one PC within the same analysis visit window, the following selection rules were applied sequentially to determine which PC was used for that time point: 1) the PC that was closer to the target date was used, 2) if PC were equal-distance in days from the target day, the later one based on measurement date and time was used, and 3) if there was more than one PC on the same day, if it was a baseline record, the largest one was used; if it was a postbaseline record, the smallest one was used.
Time Frame: Day 8 (Visit 5, EOT)
Population: Intent-to-treat population included all participants who were randomized into the study, received study medication, and had a posttreatment assessment. The ITT population was analyzed as randomized.
Measure: Mean (Standard Deviation); unit: K/mm^3
Groups:
- Cohort A: 20 mg Aavatrombopag, 1G Formulation: Participants received a 100 mg loading dose of the first generation (1G) formulation avatrombopag on Day 1, followed by 20 mg of the 1G formulation avatrombopag once daily on Days 2 to 7.
- Cohort B: 20 mg Aavatrombopag, 2G Formulation: Participants received an 80 mg loading dose of the 2G formulation avatrombopag on Day 1, followed by 20 mg 2G formulation avatrombopag once daily on Days 2 to 4 followed by 2G avatrombopag-matched placebo once daily on Days 5 to 7.
Arm/Group | Cohort A: 20 mg Aavatrombopag, 1G Formulation | Cohort A: 40 mg Avatrombopag, 1G Formulation | Cohort A: 80 mg Avatrombopag, 1G Formulation | Cohort A: Placebo, 1G Formulation | Cohort B: 10 mg Avatrombopag, 2G Formulation | Cohort B: 20 mg Aavatrombopag, 2G Formulation | Cohort B: Placebo, 2G Formulation
Number analyzed (Participants) | 18 | 16 | 17 | 16 | 21 | 21 | 21
K/mm^3 | 16.2 (10.32) | 15.9 (13.45) | 32.2 (18.59) | 3.1 (17.97) | 18.9 (10.07) | 24.9 (17.91) | 3.9 (12.49)

3. Secondary Outcome: Percentage of Participants Experiencing Dose-response by Visit
Description: as for outcome 2
Time Frame: Day 4 (Visit 3), Day 6 ( Visit 4), Day 8 (Visit 5, EOT), 3 Day Post Last Dose (Visit 6), and 7 Day Post Last Dose (Visit 7)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Groups:
- Cohort A:40 mg Avatrombopag, 1G Formulation: Participants received a 100 mg loading dose of the 1G formulation avatrombopag on Day 1, followed by 40 mg of the 1G formulation avatrombopag once daily on Days 2 to 7.
Arm/Group | Cohort A: 20 mg Avatrombopag, 1G Formulation | Cohort A:40 mg Avatrombopag, 1G Formulation | Cohort A: 80 mg Avatrombopag, 1G Formulation | Cohort A: Placebo, 1G Formulation | Cohort B: 10 mg Avatrombopag, 2G Formulation | Cohort B: 20 mg Avatrombopag, 2G Formulation | Cohort B: Placebo, 2G Formulation
Number analyzed (Participants) | 18 | 16 | 17 | 16 | 21 | 21 | 21
Percentage of participants
  Yes response (Day 4, Visit 3) | 0 | 0 | 5.9 | 0 | 0 | 4.8 | 4.8
  No response (Day 4, Visit 3) | 100.0 | 100.0 | 94.1 | 100.0 | 100.0 | 95.2 | 95.2
  Yes response (Day 6, Visit 4) | 11.1 | 12.5 | 29.4 | 0 | 14.3 | 33.3 | 9.5
  No response (Day 6, Visit 4) | 88.9 | 87.5 | 70.6 | 100.0 | 85.7 | 66.7 | 90.5
  Yes response (Day 8, Visit 5) | 38.9 | 31.3 | 76.5 | 6.3 | 42.9 | 52.4 | 9.5
  No response (Day 8, Visit 5) | 61.1 | 68.8 | 23.5 | 93.8 | 57.1 | 47.6 | 90.5
  Yes response (3 Day post last dose, Visit 6) | 55.6 | 56.3 | 82.4 | 12.5 | 66.7 | 61.9 | 9.5
  No response (3 Day post last dose, Visit 6) | 44.4 | 43.8 | 17.6 | 87.5 | 33.3 | 38.1 | 90.5
  Yes response (7 Day post last dose, Visit 7) | 61.1 | 62.5 | 88.2 | 12.5 | 71.4 | 61.9 | 9.5
  No response (7 Day post last dose, Visit 7) | 38.9 | 37.5 | 11.8 | 87.5 | 28.6 | 38.1 | 90.5

4. Secondary Outcome: Percentage of Participants Who Achieved a Platelet Count Greater Than 75,000/mm^3 on Day 4
Description: as for outcome 2
Time Frame: Day 4 (Visit 3)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Groups:
- Cohort A: 20 mg Avatrombopag, IG Formulation: Participants received a 100 mg loading dose of the first generation (1G) formulation avatrombopag on Day 1, followed by 20 mg of the 1G formulation avatrombopag once daily on Days 2 to 7.
- Cohort A: 40 mg Avatrombopag, IG Formulation: Participants received a 100 mg loading dose of the 1G formulation avatrombopag on Day 1, followed by 40 mg of the 1G formulation avatrombopag once daily on Days 2 to 7.
- Cohort A: 80 mg Avatrombopag, IG Formulation: Participants received a 100 mg loading dose of the 1G formulation avatrombopag on Day 1, followed by 80 mg of the 1G formulation avatrombopag once daily on Days 2 to 7.
- Cohort A: Placebo, IG Formulation: Participants received the 1G formulation avatrombopag-matched placebo loading dose on Day 1, then once daily on Days 2 to 7.
Arm/Group | Cohort A: 20 mg Avatrombopag, IG Formulation | Cohort A: 40 mg Avatrombopag, IG Formulation | Cohort A: 80 mg Avatrombopag, IG Formulation | Cohort A: Placebo, IG Formulation | Cohort B: 10 mg Avatrombopag, 2G Formulation | Cohort B: 20 mg Avatrombopag, 2G Formulation | Cohort B: Placebo, 2G Formulation
Number analyzed (Participants) | 18 | 16 | 17 | 16 | 21 | 21 | 21
Percentage of participants
  Yes response | 5.6 | 0 | 0 | 0 | 0 | 0 | 0
  No response | 94.4 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0

5. Secondary Outcome: Percentage of Participants Who Achieved a Platelet Count Greater Than 100,000/mm^3 on Days 4 and 8
Description: as for outcome 2
Time Frame: Day 4 (Visit 3) and Day 8 (Visit 5, EOT)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort A: 20 mg Avatrombopag, 1G Formulation | Cohort A: 40 mg Avatrombopag, 1G Formulation | Cohort A: 80 mg Avatrombopag, 1G Formulation | Cohort A: Placebo, 1G Formulation | Cohort B: 10 mg Avatrombopag, 2G Formulation | Cohort B: 20 mg Avatrombopag, 2G Formulation | Cohort B: Placebo, 2G Formulation
Number analyzed (Participants) | 18 | 16 | 17 | 16 | 21 | 21 | 21
Percentage of participants
  Yes response (Day 4, Visit 3) | 5.6 | 0 | 0 | 0 | 0 | 0 | 0
  No response (Day 4, Visit 3) | 94.4 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0
  Yes response (Day 8, Visit 5) | 5.6 | 0 | 11.8 | 0 | 4.8 | 9.5 | 0
  No response (Day 8, Visit 5) | 94.4 | 100.0 | 88.2 | 100.0 | 95.2 | 90.5 | 100.0

ADVERSE EVENTS:
Time Frame: Approximately 44 days.
Description: Treatment-emergent adverse events and treatment-emergent serious adverse events were reported. The safety population included all randomized participants who received at least one dose of study drug and had a postbaseline safety assessment. The safety population was analyzed as treated.
Arm/Group | Cohort A: 20 mg Avatrombopag, 1G Formulation | Cohort A: 40 mg Avatrombopag, 1G Formulation | Cohort A: 80 mg Avatrombopag, 1G Formulation | Cohort A: Placebo, 1G Formulation | Cohort B: 10 mg Avatrombopag, 2G Formulation | Cohort B: 20 mg Avatrombopag, 2G Formulation | Cohort B: Placebo, 2G Formulation
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/16 | 0/17 | 0/16 | 1/21 | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 3/18 | 2/16 | 3/17 | 1/16 | 5/21 | 3/21 | 3/21
Other Adverse Events (participants affected / at risk) | 17/18 | 13/16 | 13/17 | 12/16 | 17/21 | 18/21 | 16/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: 20 mg Avatrombopag, 1G Formulation (N=18) | Cohort A: 40 mg Avatrombopag, 1G Formulation (N=16) | Cohort A: 80 mg Avatrombopag, 1G Formulation (N=17) | Cohort A: Placebo, 1G Formulation (N=16) | Cohort B: 10 mg Avatrombopag, 2G Formulation (N=21) | Cohort B: 20 mg Avatrombopag, 2G Formulation (N=21) | Cohort B: Placebo, 2G Formulation (N=21)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute prerenal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Heamorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Staphylcoccal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: 20 mg Avatrombopag, 1G Formulation (N=18) | Cohort A: 40 mg Avatrombopag, 1G Formulation (N=16) | Cohort A: 80 mg Avatrombopag, 1G Formulation (N=17) | Cohort A: Placebo, 1G Formulation (N=16) | Cohort B: 10 mg Avatrombopag, 2G Formulation (N=21) | Cohort B: 20 mg Avatrombopag, 2G Formulation (N=21) | Cohort B: Placebo, 2G Formulation (N=21)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiomegaly (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 2 | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 4 | 1 | 1 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 3
Colonic polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 0 | 3 | 2
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 1
Erosive duodenitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastric polyps (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 0
Gastric verices (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 2 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 2 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 2 | 2 | 5 | 2 | 3
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Oesophageal mass (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Polyp colorectal (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Portal hypertensive gastropathy (Gastrointestinal disorders) | 4 | 2 | 0 | 0 | 3 | 0 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Varices oesophageal (Gastrointestinal disorders) | 2 | 2 | 0 | 1 | 1 | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 3 | 0 | 0 | 1 | 1
Chills (General disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0
Fatigue (General disorders) | 4 | 1 | 0 | 1 | 2 | 2 | 4
Hyperthermia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Irritability (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 2 | 0 | 2 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 2 | 2 | 1 | 0 | 3
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 2 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Fungal skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Helicobacter infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitus (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Staphylococcal skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthropid bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Iris injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 2 | 2 | 0 | 1 | 1 | 2
Scratch (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Blood glucose increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood urine present (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram T wave peaked (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Glucose urine present (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Heart rate increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urine output decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0 | 2 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 1 | 1 | 3 | 1 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 1 | 2 | 1 | 3 | 3
Hepatic encephalopathy (Nervous system disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Unresponsive to stimuli (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 1
Listless (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Mental status change (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute prerenal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Scrotal swelling (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pulmonary valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Ocular icterus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Faeces discolored (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Aortic arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other